CLINICAL TRIAL: NCT03461900
Title: Guided Fluid-balance Optimization With Mini-fluid chALlenge During Septic Shock: A Multicenter, Stepped Wedge Cluster Randomized Trial
Brief Title: Guided Fluid-balance Optimization With Mini-fluid chALlenge During Septic Shock
Acronym: GOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29BRC18.0054
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-03

CONDITIONS: Septic Shock
Keywords: Septic shock; Fluid optimisation; Minifluid challenge; Fluid overload
MeSH Terms: conditions — Shock, Septic; Edema

STUDY DESIGN:
Intervention Model Description: stepped wedge cluster randomized trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Minifluid challenge (Experimental): 100 ml of 4% Albumin will be deliver to assess fluid responsiveness
  Interventions: Other: Minifluid challenge
- Control (Experimental): Patient will be treated as defined by most recent surviving sepsis campaign guidelines
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: Minifluid challenge — Pragmatic optimization fluid management protocol based on Mini-Fluid Challenge (MFC) in treating an acute circulatory failure. MFC consist of an infusion of 100 ml of colloid solution (4% human serum albumin) during 1 minute via a separate venous line. Before and after each MFC and depending on the hemodynamic device used, the attending physician will perform a first set of hemodynamic measurements, including cardiac index (CI) or cardiac output (CO); stroke volume (SV), indexed stroke volume (iSV) or velocity time index (VTI). If the variation in measurement is superior to 10%, the attending physician will infuse 400 ml of buffered crystalloid solution or saline solution. After an infusion of 500 ml, fluid responsiveness will be evaluated with CI or CO measurement. For non-responders, fluid challenge must be stopped and other therapeutics should be considered. For responder, another MFC should be consider if hemodynamic status is not stabilized.
  Arms: Minifluid challenge
Other: Usual practice — Patients included in control group will be managed according to the last surviving sepsis recommendations edited in 2017.
  Arms: Control

SUMMARY:
Many observational studies have highlighted an independent association between fluid overload and clinical outcomes during septic shock. To optimize fluid balance, clinician has several options to consider carefully fluid administration and avoid fluid overload. More than a general restrictive approach, a pragmatic, individual tailored approach should be considered to optimize patients' hemodynamics during acute circulatory failure. Many advances in hemodynamic monitoring were described. Mini-fluid challenge appears to be a sensible method to use for bedside assessment to optimize fluid infusion. The next step for hemodynamic management in the ICU should be to test a hemodynamic goal-directed approach to better control fluid management and eventually improve patient's outcome. The main objective of the GOAL study is to evaluate a pragmatic optimization fluid management protocol tailored to each patient's hemodynamic status based on mini-fluid challenges. This intervention will be compared to usual management based on the latest guidelines. This intervention aims to decrease organ dysfunction during septic shock. This is the first large clinical trial designed to test this hypothesis.

DETAILED DESCRIPTION:
GOAL study is a stepped wedge cluster-randomized trial. Centers will switch randomly from the control to the intervention at regular intervals:

* Control periods: Patients receive a usual optimization fluid management according to surviving sepsis campaign guidelines.
* Interventional periods: Patients receive a pragmatic, protocolized and individual optimization fluid management according to validated components of a hemodynamic challenges called Mini-Fluid Challenge (MFC).

Except fluid therapy in interventional group, management of sepsis will be at the discretion of the attending physician. The use of international guidelines for all therapeutic interventions is recommended in all patients whenever their group.

All patients will be followed from enrolment to death or hospital discharge. If alive but not in the hospital after 28 days since septic shock, clinical outcomes will be evaluated by a visit with an intensivist or, if a physical examination is not possible, by a telephone interview performed by an intensivist. To ensure the same data collection in all centers, visits were planned: D0 (inclusion), D1 to D10 (in ICUs), D28 and D180.

Classical blinded methods cannot be used in case of evaluation of an optimization protocol. Investigators are unblinded to which arm patient is randomized. To ensure the same evaluation for all patients and in all centers, all events recorded will be evaluated by an independent clinical event committee.

All primary endpoints will be analyzed according to a hierarchized analysis to ensure comparison of multiple issues without considering type I error inflation. Secondary outcomes will be analyzed as exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (Age > 18 years)
* Admitted in ICU for less than 3 days.
* Abdominal (excepted urinary tract infection) or pulmonary related septic shock, defined by SEPSIS III criteria diagnosed within less than 12 hours.
* Written consent or oral by the patient (and/or consent signed by the next of skin)
* Patient has social security affiliation or who beneficiary of such social security

Exclusion Criteria:

* Patient with life expectancy inferior to 24 hours at the time of inclusion.
* Cardiac arrest
* Allergy to albumin
* Pregnancy
* Traumatic brain injury
* Limitation of invasive therapeutics, palliative care
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Delta SOFA score (Day0 - Day5) | Day 5
  Delta SOFA score is the difference between SOFA (Sepsis-related Organ Failure Assessment) measured at day 0 and at Day 5. SOFA score was developed to quantify organ dysfunction in patients with sepsis and to determine treatment effectiveness. SOFA score is a scale range from 0 to 24, with higher scores indicating worse organ dysfunction. Five organs dysfunctions are analyzed:
  * Respiratory: PaO2/FiO2 ratio
  * Cardio-vascular: severity of hypotension and need of vasopressors (µ/kg/min)
  * Renal: creatinine (mg/dl)
  * Hemostasis: Platelet count (G/l)
  * Liver: Bilirubin (mg/dl)
  * Neurologic: Glasgow coma scale
ICU length of stay until ability to ICU discharge | 90 days
Length of stay in hospital | 90 days
Ventilator free days at day 28 | 28 days
Renal failure free days at day 28 | 28 days
Catecholamine free days at day 10 | 10 days

SECONDARY OUTCOMES:
Mortality at day 28 | 28 days
Mortality at day 90 | 90 days

OTHER OUTCOMES:
SF-36 (Short-Form 36) | 6 months
  The SF-36 is an indicator of health status and quality of life. The SF-36 has eight dimensions; the scores are weighted sums of the questions in each section. This scores range from 0 - 100. Lower scores indicate more disability and higher scores less disability.
  The eight dimensions of this score are:
  * Vitality
  * Physical functioning
  * Bodily pain
  * General health perceptions
  * Physical role functioning
  * Emotional role functioning
  * Social role functioning
  * Mental health
CANTAB test (Cambridge Neuropsychological Test Automated Battery) | 6 months
  CANTAB test have demonstrated sensitivity to detecting changes in neuropsychological performance and include tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control
PCL-5 | 6 months
  Quality of life with PCL-5 questionnaire

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Angers university hospital, Angers
  - Besançon university hospital, Besançon
  - Brest university hospital, Brest
  - Chartres Hospital, Chartres
  - Clermont Ferrand university hospital, Clermont-Ferrand
  - Le Mans hospital, Le Mans
  - Marseille university horpital, Marseille
  - Morlaix hospital, Morlaix
  - Nantes university hospital, Nantes
  - Nîmes university hospital, Nîmes
  - George Pompidou university hospital (APHP), Paris
  - Kremlin Bicêtre university hospital (APHP), Paris
  - Poitiers university hospital, Poitiers
  - Rouen university hospital, Rouen
  - Toulon hospital, Toulon
  - Tours university hospital, Tours
  - Hôpital privé de l'ouest parisen, Trappes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: All collected data that underlie results in a publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Malbrain ML, Marik PE, Witters I, Cordemans C, Kirkpatrick AW, Roberts DJ, Van Regenmortel N. Fluid overload, de-resuscitation, and outcomes in critically ill or injured patients: a systematic review with suggestions for clinical practice. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):361-80. doi: 10.5603/AIT.2014.0060. PMID 25432556
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Sakr Y, Rubatto Birri PN, Kotfis K, Nanchal R, Shah B, Kluge S, Schroeder ME, Marshall JC, Vincent JL; Intensive Care Over Nations Investigators. Higher Fluid Balance Increases the Risk of Death From Sepsis: Results From a Large International Audit. Crit Care Med. 2017 Mar;45(3):386-394. doi: 10.1097/CCM.0000000000002189. PMID 27922878
- [Background] Marik PE, Linde-Zwirble WT, Bittner EA, Sahatjian J, Hansell D. Fluid administration in severe sepsis and septic shock, patterns and outcomes: an analysis of a large national database. Intensive Care Med. 2017 May;43(5):625-632. doi: 10.1007/s00134-016-4675-y. Epub 2017 Jan 27. PMID 28130687
- [Background] Cecconi M, Hofer C, Teboul JL, Pettila V, Wilkman E, Molnar Z, Della Rocca G, Aldecoa C, Artigas A, Jog S, Sander M, Spies C, Lefrant JY, De Backer D; FENICE Investigators; ESICM Trial Group. Fluid challenges in intensive care: the FENICE study: A global inception cohort study. Intensive Care Med. 2015 Sep;41(9):1529-37. doi: 10.1007/s00134-015-3850-x. Epub 2015 Jul 11. PMID 26162676